CLINICAL TRIAL: NCT00102063
Title: Aripiprazole in Adolescents With Schizophrenia
Acronym: APEX 239
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31-03-239
Record Dates: First submitted 2005-01-19; First posted 2005-01-20 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Aripiprazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Aripiprazole 10 mg/day Group (Active Comparator): Dose was titrated to a target dose of 10 mg/day as follows: starting dose 2 mg/day, increased to 5 mg/day on Day 3, 10 mg/day on Day 5; one dose reduction to 5 mg/day allowed after Day 25
  Interventions: Drug: Aripiprazole tablet, 10 mg
- Aripiprazole 30 mg/day Group (Active Comparator): Dose was titrated to a target dose of 30 mg/day as follows: starting dose 2 mg/day, increased to 5 mg/day on Day 3, 10 mg/day on Day 5, 15 mg/day on Day 7, 20 mg/day on Day 9, and 30 mg/day on Day 11; one dose reduction to 15 mg/day allowed after Day 25
  Interventions: Drug: Aripiprazole tablet, 30 mg
- Placebo Group (Placebo Comparator): Participants were given a single pill administered once daily
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Aripiprazole tablet, 10 mg — Aripiprazole tablet 10 mg po qd x 42 days
  Other Names: OPC-14597
  Arms: Aripiprazole 10 mg/day Group
Drug: Aripiprazole tablet, 30 mg — Aripiprazole tablet 30 mg po qd x 42 days
  Other Names: OPC-14597
  Arms: Aripiprazole 30 mg/day Group
Drug: Placebo tablet — Placebo tablet po qd x 42 days
  Arms: Placebo Group

SUMMARY:
The purpose of this trial is to test the safety and efficacy of aripiprazole in adolescent patients with schizophrenia for a period of at least 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Schizophrenia 1

Exclusion Criteria:

* Patients diagnosed with schizoaffective disorder, major depressive disorder, delirium, or bipolar disorder

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2004-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaretta Nyilas, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (55):
- United States (53):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Costa Mesa, California
  - Local Institution, Los Angeles, California
  - Local Institution, National City, California
  - Local Institution, Orange, California
  - Local Institution, Pasadena, California
  - Local Institution, Sacramento, California
  - Local Institution, San Diego, California
  - Local Institution, Temecula, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Gainesville, Florida
  - Local Institution, Hialeah, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, North Miami, Florida
  - Local Institution, Orange City, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Newnan, Georgia
  - Local Institution, Smyrna, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Kansas City, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Lake Charles, Louisiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Medford, Massachusetts
  - Local Institution, Clinton Township, Michigan
  - Local Institution, Flowood, Mississippi
  - Local Institution, Kansas City, Missouri
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Elmsford, New York
  - Local Institution, New York, New York
  - Local Institution, Olean, New York
  - Local Institution, Rochester, New York
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Cleveland, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Bala-Cynwyd, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Memphis, Tennessee
  - Local Institution, Bellaire, Texas
  - Local Institution, DeSoto, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Richmond, Virginia
  - Local Institution, Kirkland, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Wauwatosa, Wisconsin
- Puerto Rico (2):
  - Local Institution, Rio Piedras
  - Local Institution, San Juan

REFERENCES:
- [Derived] Correll CU, Zhao J, Carson W, Marcus R, McQuade R, Forbes RA, Mankoski R. Early antipsychotic response to aripiprazole in adolescents with schizophrenia: predictive value for clinical outcomes. J Am Acad Child Adolesc Psychiatry. 2013 Jul;52(7):689-698.e3. doi: 10.1016/j.jaac.2013.04.018. Epub 2013 Jun 5. PMID 23800482
- [Derived] Robb AS, Carson WH, Nyilas M, Ali M, Forbes RA, Iwamoto T, Assuncao-Talbott S, Whitehead R, Pikalov A. Changes in positive and negative syndrome scale-derived hostility factor in adolescents with schizophrenia treated with aripiprazole: post hoc analysis of randomized clinical trial data. J Child Adolesc Psychopharmacol. 2010 Feb;20(1):33-8. doi: 10.1089/cap.2008.0163. PMID 20166794
- [Derived] Findling RL, Robb A, Nyilas M, Forbes RA, Jin N, Ivanova S, Marcus R, McQuade RD, Iwamoto T, Carson WH. A multiple-center, randomized, double-blind, placebo-controlled study of oral aripiprazole for treatment of adolescents with schizophrenia. Am J Psychiatry. 2008 Nov;165(11):1432-41. doi: 10.1176/appi.ajp.2008.07061035. Epub 2008 Sep 2. PMID 18765484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 101 centers in the United States, Europe, South America, the Caribbean, and South Africa between August 2004 and August 2006.
Pre-assignment Details: Participants were screened over a 4-week period.
Period: Overall Study
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Started | 100 | 102 | 100
Completed | 84 | 84 | 90
Not Completed | 16 | 18 | 10
Not completed — Lack of Efficacy | 5 | 1 | 1
Not completed — Adverse Event | 7 | 4 | 2
Not completed — Withdrawal by Subject | 4 | 12 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group | Total
Number analyzed (Participants) | 100 | 102 | 100 | 302
Age Continuous [Mean (Standard Deviation); unit: years] | 15.6 (1.3) | 15.4 (1.4) | 15.4 (1.4) | 15.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 37 | 39 | 131
  Male | 45 | 65 | 61 | 171
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 16 | 12 | 15 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 11 | 6 | 34
  White | 54 | 62 | 64 | 180
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 17 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: Change from baseline to last observed post-baseline value in PANSS total score, using the last observation carried forward.
  This scale consists of symptom constructs (7 positive, 7 negative, 16 general psychopathology), each to be rated on a 7-point scale of severity with 1 being absent to 7 being extreme. Minimum score is 30 which is best outcome; maximum score is 210 for worse outcome.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Error); unit: points
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 99 | 97 | 98
points | -26.7 (1.9) | -28.6 (0.9) | -21.2 (1.9)
Statistical Analysis 1: Comparison: Aripiprazole 10 mg/Day Group vs Placebo Group; Test type: Superiority or Other; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Aripiprazole 30 mg/Day Group vs Placebo Group; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

2. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Positive Subscale Score
Description: Change from baseline to last observed post-baseline value in PANSS positive subscale score, using the last observation carried forward.
  Scale consists of 7 positive symptom constructs each to be rated on a 7- point scale of severity with 1 = absent to 7 = extreme. Minimum score is 7 which is best outcome; maximum score is 49 for worse outcome.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Error); unit: points
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 98 | 99 | 97
points | -7.6 (0.6) | -8.1 (0.6) | -5.6 (0.6)

3. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Negative Subscale Score
Description: Change from baseline to last observed post-baseline value in PANSS Negative Subscale score, using the last observation carried forward.
  Scale consists of 7 negative symptom constructs each to be rated on a 7- point scale of severity with 1 = absent to 7 = extreme. Minimum score is 7 which is best outcome; maximum score is 49 for worse outcome.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Error); unit: points
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 99 | 97 | 98
points | -6.9 (0.6) | -6.6 (0.6) | -5.4 (0.6)

4. Secondary Outcome: Change in Clinical Global Impression (CGI) Severity Score
Description: Change from baseline to last observed post-baseline value in CGI severity score, using the last observation carried forward.
  Scale refers to the global impression of the subject with respect to severity of the illness. The scale rates the subject's severity of illness from 0 (not rated) to 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Day 42
Measure: Mean (Standard Error); unit: points
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 99 | 97 | 98
points | -1.2 (0.1) | -1.3 (0.1) | -0.9 (0.1)

5. Secondary Outcome: Clinical Global Impression (CGI) Improvement Score
Description: Last observed post-baseline value in CGI improvement score, using the last observation carried forward.
  Scale refers to the global impression of the subject with respect to improvement of the illness. The scale rates the subject's severity of illness from 0 (not rated) to 1 (least severe) to 7 (most severe).
Time Frame: Baseline and Day 42
Measure: Mean (Standard Error); unit: points
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 99 | 97 | 98
points | 2.7 (0.1) | 2.5 (0.1) | 3.1 (0.1)

6. Secondary Outcome: Change in Children's Global Assessment Scale (CGAS) Score
Description: Change from baseline to last observed post-baseline value in CGAS score, using the last observation carried forward.
  Scale is a 100-point scale measuring psychological, social, and school functioning for children aged 6 to 17 years. Minimum scores ranged from 1-10, representing the need for constant supervision (worse outcome) to maximum scores of 91-100, representing superior functioning (better outcome).
Time Frame: Baseline and Day 42
Measure: Mean (Standard Error); unit: points
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 99 | 97 | 98
points | 14.7 (1.5) | 14.8 (1.3) | 9.8 (1.3)

7. Other Pre Specified Outcome: Change in Pediatric Quality of Life Enjoyment and Satisfaction (PQLES) Questionnaire Total Score
Description: Change from baseline to last observed post-baseline value in PQLES total score, using the last observation carried forward.
  Scale consists of 14 items pertaining to daily life activities and satisfaction, and an overall assessment item. Each item will be rated on a five-point scale (1=very poor, 2=poor, 3=fair, 4=good, 5=very good) with a minimum score of 14 (better outcome) and a maximum score of 70 (worse outcome).
Time Frame: Baseline and Day 42
Measure: Mean (Standard Error); unit: points
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 99 | 97 | 98
points | 5.2 (0.9) | 5.9 (0.9) | 4.5 (0.9)

8. Other Pre Specified Outcome: Patients Achieving Remission
Description: The number of subjects achieving remission. Remission was defined as a score of mild or less (≤ 3) for items P1, P2, P3, N1, N4, N6, G5, and G9 in the PANSS score.
Time Frame: Baseline and Day 42
Measure: Number; unit: participants
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Number analyzed (Participants) | 99 | 97 | 98
participants | 53 | 56 | 35

ADVERSE EVENTS:
Time Frame: Adverse event data were collected as spontaneous reports at all scheduled visits. Serious AEs were monitored until the subject's health returned to baseline status or other parameters returned to normal or were otherwise explained.
Arm/Group | Aripiprazole 10 mg/Day Group | Aripiprazole 30 mg/Day Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 4/100 | 4/102 | 3/100
Other Adverse Events (participants affected / at risk) | 71/100 | 74/102 | 57/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 10 mg/Day Group (N=100) | Aripiprazole 30 mg/Day Group (N=102) | Placebo Group (N=100)
Varicella (Infections and infestations) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 1 | 0 | 0 — Event did not meet the criteria for neuroleptic syndrome
Aggression (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 1
Schizophrenia (Psychiatric disorders) | 1 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 10 mg/Day Group (N=100) | Aripiprazole 30 mg/Day Group (N=102) | Placebo Group (N=100)
Nausea (Gastrointestinal disorders) | 9 | 10 | 6
Vomiting (Gastrointestinal disorders) | 5 | 3 | 5
Nasopharyngitis (Infections and infestations) | 5 | 5 | 4
Akathisia (Nervous system disorders) | 5 | 5 | 12
Dizziness (Nervous system disorders) | 7 | 4 | 3
Extrapyramidal disorder (Nervous system disorders) | 13 | 22 | 5
Headache (Nervous system disorders) | 16 | 11 | 10
Somnolence (Nervous system disorders) | 11 | 22 | 6
Tremor (Nervous system disorders) | 2 | 12 | 2
Agitation (Psychiatric disorders) | 1 | 3 | 5
Insomnia (Psychiatric disorders) | 11 | 10 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No